CLINICAL TRIAL: NCT01926054
Title: An Open Label Randomized Phase IV Study of the Safety and Efficacy of ACTHAR GEL in Patients With Membranous (Class V) Lupus Nephritis
Brief Title: ACTHAR GEL in Patients With Membranous (Class V) Lupus Nephritis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Ohio State University (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Brad Rovin, MD, Principle Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013H0121
Record Dates: First submitted 2013-07-15; First posted 2013-08-20 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: SLE Glomerulonephritis Syndrome, WHO Class V
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acthar Gel 80 IU SC BIW (Active Comparator): 80 IU administered subcutaneously BIW for 6 months
  Interventions: Drug: Acthar gel
- Acthar Gel 80 IU SC TIW (Active Comparator): 80 IU administered subcutaneously TIW for 6 months
  Interventions: Drug: Acthar gel

INTERVENTIONS:
Drug: Acthar gel

SUMMARY:
This is an open-label, randomized, multi-center, Phase IV study of Acthar Gel in patients with biopsy-proven membranous (Class V) lupus nephritis (LN) aimed at providing proof-of-concept data that Acthar is a safe and effective therapy for membranous LN. Class V LN is a secondary form of membranous nephropathy, and occurs in 8-20% of patients with LN.

Two different doses of Acthar Gel will be tested. The active intervention phase of this study will take place over 6 months, and follow-up will occur over the following 6 months. Efficacy and safety of the use of Acthar Gel for treatment of membranous LN will be assessed and analyzed throughout the course of the study by laboratory testing, physical exams, and other evaluation tools. Subjects will be closely monitored for adverse effects associated with the use of Acthar gel and if necessary study drug dosing will be reduced. The anticipated benefits to subjects are a complete renal response rate of 40% at 6 months showing superiority over the published complete remission rates of the currently used immunosuppressive therapies, and no unexpected toxicity signals.

Pure Class V LN affects a significant number of systemic lupus erythematosus (SLE) patients and although it is less aggressive than proliferative forms of LN it still causes important renal and non-renal morbidity and mortality over time, especially in patients who remain nephrotic. The therapy of Class V LN is not clear, and currently used therapies are highly toxic because of immunosuppression, risk of infertility, and risk of future malignancy. Additionally, these therapies are only modestly effective in inducing remissions of Class V LN. There is thus an unmet need for a more effective and less toxic treatment for Class V LN.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age who have pure Class V LN or Class V+II LN diagnosed by a kidney biopsy within 4 months of screening. If a patient has segmental glomerular scarring indicative of previous Class III or IV lesions, but no evidence of current Class III or IV activity, and only the Class V component is active, they can be enrolled, despite having a mandatory ISN/RPA classification of Class V + III or IV
* Proteinuria ≥ 3 g/d despite adequate blood pressure control defined as systolic blood pressure ≤ 130 mm Hg 75% of the time, per the clinical judgment of the site investigator.
* Serum creatinine < 2 mg/dl or eGFR > 30 ml/minute

Exclusion Criteria:

* Patients < 18 years of age

  * Pregnancy or planning to become pregnant anytime throughout their participation in the trial, up until 30 days after last dose of study drug.
  * Kidney biopsy with active Class III or IV LN
  * More than 50% interstitial fibrosis and/or glomerulosclerosis on kidney biopsy
  * Patients with hepatitis B, C, HIV, TB or other active and chronic infections at the time of screening
  * Patients with liver disease and transaminases greater than 2.5 times the upper limit of normal of the laboratory, patients with diabetes mellitus type I or II, patients with refractory hypokalemia, patients with Cushing's Disease or Syndrome
  * Patients who have been treated with cyclophosphamide, cyclosporine A, tacrolimus, B-cell depleting therapies, or experimental therapies including biologics within 6 months of screening
  * Patients with active neuropsychiatric lupus, lupus pneumonitis, lupus vasculitis at screening
  * Patients with high or very high extra-renal lupus activity defined as an xSLEDAI score greater than 10 at the time of screening
  * Patients who have received high-dose intravenous methylprednisolone (1 g cumulative) within 3 months of screening
  * Patients currently receiving, or who have received MMF or AZA in the 3 months preceding enrollment for extra-renal SLE.
  * Patients who have received methotrexate or who are receiving methotrexate and it can be discontinued will be eligible; if methotrexate cannot be stopped safely, the patient will not be eligible.
  * Patients currently receiving more than 20 mg/d prednisone that cannot be safely reduced to 20mg/d or less beginning at least one month before enrollment on day 0
  * Patients who are not on a stable dose of Anti-Malarials and/or Anti-hypertensives at least one month preceding baseline visit and during the study. (Refer to allowed medication section)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2018-02 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Baseline and Month 12
  Measuring adverse events and serious adverse events taking Acthar Gel in Class V lupus nephritis
Change in laboratory data | Baseline and Month 12
  changes in laboratory parameters, and metabolic side effects such as hyperglycemia, hypokalemia, and hyperlipidemia
Renal Response to Acthar Gel | Baseline and Month 6
  Change in Proteinuria and serum creatinine

SECONDARY OUTCOMES:
Change in remission | Month 6 and Month 12
  To determine the duration of complete and partial remission after study drug is stopped
Change baseline SLE laboratory | Baseline and month 6
  To determine the effect of Acthar Gel on baseline levels of anti-double stranded DNA (dsDNA) antibodies and complement components C3 and C4
Change in extra-renal systemic lupus erythematosus disease activity index | Baseline and Month 6
  To determine the effect of Acthar Gel on the patients global assessment score, the physicians global assessments score and xSLEDAI

OTHER OUTCOMES:
reduction of urine protein to creatinine ratio | week 8 and month 6
  To determine if a reduction of the urine protein-to-creatinine ratio (uPCR) of an intended 24-hour of ≥25% at 8 weeks predicts complete or partial response at 6 months
change urine monocyte chemotactic protein-1 and urine vascular endothelial growth factor | Baseline and 6 month
  To determine change from baseline of urine monocyte chemotactic protein-1 (uMCP1) and urine vascular endothelial growth factor (uVEGF) at 3 and 6 months
percent of patients who have renal and non renal flares | baseline and month 12
  To determine the % of patients who have renal flares during treatment and during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Brad H Rovin, MD, Principal Investigator — The Ohio State University Wexner Medical Center, Division of Nephrology
Locations (1):
- The Ohio State University Wexner Medical Center, Nephrology Clinical Trials Unit, Columbus, Ohio, United States